CLINICAL TRIAL: NCT06445205
Title: Utilising Volumetric Absorptive Microsampling (VAMS®) Technology to Monitor Tacrolimus and Creatinine Concentrations in Adult Renal Transplant Patients
Brief Title: Utilising Volumetric Absorptive Microsampling (VAMS) Technology to Monitor Tacrolimus and Creatinine
Status: Suspended | Type: Observational
Why Stopped: Chief Investigator not available
Sponsor: Lancashire Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 322562; 22/PR/1599 (Other: Health research Authority)
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2024-05

CONDITIONS: Kidney Transplant Rejection; Kidney Replacement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sample collection: Sample collection via standard phlebotomy as well as point-or-care Mitra device.
  Interventions: Diagnostic Test: Mitra® device with VAMS® (volumetric absorptive microsampling) technology

INTERVENTIONS:
Diagnostic Test: Mitra® device with VAMS® (volumetric absorptive microsampling) technology — Capillary blood sample

SUMMARY:
Tacrolimus is a medicine given to try and stop rejection of a new kidney after transplant surgery. If too much taken the kidney may be damaged. If not enough taken, the risk of rejection is increased. Creatinine is a waste product made by the muscles and is normally removed from the body by the kidneys. If kidney function gets worse, the creatinine level in the blood goes up and means the new new kidney is not working properly. It is important to monitor levels of tacrolimus and creatinine regularly, to keep the kidney as healthy as possible. Regular monitoring also aids with balancing the amount of tacrolimus that patients need to take.

The COVID-19 pandemic led to changes in the delivery of transplant services. One such changes was a move to the use of point-of-care, and at home devices.

The study involves the set-up a new method in an NHS laboratory to test tacrolimus and creatinine levels in blood collected in the normal blood tubes and to compare the results with this new collection device, to see if the results are the same.

If the results match, patients will continue to collect a blood sample using the new devices and send it to the laboratory. This will save both patients and the NHS time and money as they will not have to travel to a hospital to have their bloods taken.

DETAILED DESCRIPTION:
A minimum of 50 adult renal transplant patients (>18 years old) taking tacrolimus as an immunosuppressant will be recruited when attending their routine outpatient follow up appointment, or if selected as eligible by the Renal Consultants and transplant nurses. Written consent will be obtained from all participants.

Patients attending blood clinic to have their routine blood samples taken will also have a finger prick and a small amount of blood (10µl) will be collected by volumetric absorptive micro sampling (VAMS) using the Mitra® device (Neoteryx), according to manufacturer's instructions. Two venous blood samples will be collected from the patients by venepuncture by trained phlebotomists/nurses. A 4ml EDTA and a 4ml serum gel sample (to measure tacrolimus and renal function as part of routine care). Tacrolimus and creatinine are measured in venous blood samples as part of routine patient care therefore these will be processed as normal, and results reported. The paired capillary samples collected using the Mitra® device will be batched and run when appropriate by liquid chromatography-mass spectrometry (LC-MS/MS). Mitra® devices will be stored at -20 degree Celsius, prior to analysis.

Venous EDTA whole blood samples (collected by venepuncture) and capillary whole blood samples (collected by VAMS®) will be analysed for tacrolimus using a validated LC-MS/MS assay in routine clinical use in the lab using the Waters ACQUITY UPLC system and Xevo TQD MS. Capillary whole blood samples (collected by VAMS®) and serum samples will be analysed for creatinine using an LC-MS/MS method which will be developed in house. For the method comparison, serum samples (collected by venepuncture) will be analysed for creatinine using an enzymatic method on the Roche platform. All sample analysis will be performed in an ISO 15189 accredited laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Post renal transplant patients taking tacrolimus
* having regular bloods taken for tacrolimus and renal function testing.
* Patients must be taking tacrolimus as part of their immunosuppressive regimen.
* They must be over 18 years of age

Exclusion Criteria:

* Patients under the age of 18 (the study is for adults only).
* Vulnerable adults who are deemed unable to give consent themselves - If applicable, this can be assessed using the Trust clinical tool 'Assessment of Mental Capacity'.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult renal transplant patients (>18 years old) taking tacrolimus as an immunosuppressant
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Tacrolimus in Capillary Blood Samples | 6 months
  That Tacrolimus is within range: 10-20ng/ml
Creatinine in Capillary Blood Samples | 6 months
  That Creatinine is within range: 52.2 - 119.3 micromoles/L

SECONDARY OUTCOMES:
Tacrolimus is concordant with venous blood sample | 6 months
  Results match standard venous results for Tacrolimus and is within range:10-20ng/ml then use of VAMS will be implemented into routine clinical practice for monitoring renal patients post transplant.
Creatinine is concordant with venous blood sample | 6 months
  Results match standard venous results for Creatinine and is within range: 52.2 - 119.3 micromoles/L.

CONTACTS AND LOCATIONS:
Overall Officials: Kina Bennett, PhD, Study Chair — Lancashire Teaching Hospitals NHS Foundation Trust
Locations (1):
- Lancashire Teaching Hospitals NHS Foundation Trust, Preston, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-01-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT06445205/Prot_000.pdf